CLINICAL TRIAL: NCT03314675
Title: Assessment of Pacing Stimulus Conduction and Latency Measurements in CRT-D Patients
Acronym: BIO|PULSE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unsuccessful enrollment
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CR022
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Heart Failure
Keywords: CRT-D, LV Latency
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CRT-D Measurements (Other): Pre-specified measurements and additional follow-ups
  Interventions: Device: BIOTRONIK CRT-D

INTERVENTIONS:
Device: BIOTRONIK CRT-D — Pre-specified follow-up and measurements

SUMMARY:
The study is designed to collect data on LV latency in CRT-D patients by the CRT-D and compare measurements to 12-lead ECG data

ELIGIBILITY:
Inclusion Criteria:

* Patient has been implanted with a CRT-D device by BIOTRONIK at least 4 weeks before enrollment date
* Patient successfully implanted with a left ventricular lead
* High likelihood of LV latency ≥ 40 ms
* LV lead in lateral or postero-lateral position in the coronary venous system
* Patient is able to understand the nature of the clinical investigation
* Patient is willing to undergo the required measurements at the investigation site
* Patient provides written informed consent
* Age ≥ 18 years

Exclusion Criteria:

* Patients with irregular ventricular rhythm due to atrial tachycardia
* Pregnant or breast-feeding women
* Participation in an interventional clinical investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
Rate of patients with LV latency >/= 40ms (stimulus to QRS onset) with respect to the total number of screened patients | 1 day

SECONDARY OUTCOMES:
Device-base measured LV latency in the LV IEGM channel and Far Field channel | 1 day
12-lead ECG-measured LV latency in the channel with earliest QRS onset | 1 day
Device-based measured latency intervals (stimulus to electrogram peak and end) in the LV IEGM channel and the Far Field channel | 1 day
12-lead ECG-measured latency intervals | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nordbeck, PD Dr., Principal Investigator — Wuerzburg University Hospital
Locations (7):
- Czechia (2):
  - Ceske Budejovice hospital, České Budějovice
  - Institute for Clinical and Experimental Medicine, Prague
- Germany (4):
  - Herz- und Diabetiszentrum NRW, Bad Oeynhausen
  - SRH Waldklinikum Gera GmbH, Gera
  - Universitätsklinikum Gießen und Marburg, Giessen
  - Universitätsklinikum Würzburg, Würzburg
- The Erasmus University Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No